CLINICAL TRIAL: NCT00138047
Title: Randomized, Double-Blind, Placebo-Controlled Trial of Zinc Supplementation in HIV-1-Infected Children
Brief Title: Safety and Efficacy of Zinc Supplementation in HIV-1-Infected Children in South Africa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); University of KwaZulu (Other); Grey's Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H.22.02.03.25.B1
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2005-12-05 (Estimated); Status verified 2005-08

CONDITIONS: HIV Infections
Keywords: zinc; HIV; children
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: zinc supplementation

SUMMARY:
The goal of the study is to rule out a harmful effect of zinc supplementation in HIV-1-infected children. The null hypothesis is that zinc supplementation will increase plasma HIV RNA levels.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled equivalence trial of zinc supplementation was conducted at Grey's Hospital in Pietermaritzburg, South Africa. Ninety-six HIV-1-infected children were randomly assigned to receive 10 mg of elemental zinc as sulfate or placebo daily for 6 months. Baseline measurements of plasma HIV-1 viral load and the percentage of CD4+ T-lymphocytes were established at two study visits prior to randomization, and measurements were repeated 3, 6 and 9 months after starting supplementation. Plasma HIV-1 viral load and the percentage of CD4+ T-lymphocytes were compared before and after supplementation.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection
* 6 to 60 months of age
* Not receiving antiretroviral therapy
* Cared for as outpatients at Grey's Hospital

Exclusion Criteria:

* Receiving antiretroviral therapy

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2003-03; Study Completion 2004-09

PRIMARY OUTCOMES:
mean difference in log10 HIV-1 viral load at each visit

SECONDARY OUTCOMES:
mean difference in percentage of CD4+ T-cells at each visit
number of illness visits

CONTACTS AND LOCATIONS:
Overall Officials: William J Moss, MD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Robert E Black, MD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Raziya Bobat, MBChB, MD, Principal Investigator — Nelson R Mandela School of Medicine, University of KwaZulu-Natal; Hoosen Coovadia, MD, MBBS, Principal Investigator — Doris Duke Medical Research Institute, University of KwaZulu-Natal
Locations (1):
- Grey's Hospital, Pietermaritzburg, South Africa